CLINICAL TRIAL: NCT03237806
Title: Effects of Sedation on Transpulmonary Pressure and Lung Homogenous of ARDS Patients
Brief Title: Effects of Sedation on Transpulmonary Pressure and Lung Homogenous
Acronym: ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2012ZDIIKY22.0
Record Dates: First submitted 2014-05-21; First posted 2017-08-03 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: ARDS
Keywords: ARDS,; Transpulmonary pressure,; Sedation
MeSH Terms: interventions — Deep Sedation

STUDY DESIGN:
Intervention Model Description: Self control
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baseline (No Intervention): In this phase, patients were sedated to the level of Ramsay 6 before Deep sedated or Light sedated
- Deep sedation (Experimental): In this Arm, patients were sedated to the level of Ramsay 5(Deep sedated) by Midazolam IV continuously
  Interventions: Drug: Deep sedated
- Light sedation (Experimental): In this Arm, patients were sedated to the level of Ramsay 3(Light sedated)by Midazolam IV continuously
  Interventions: Drug: Light sedated

INTERVENTIONS:
Drug: Deep sedated — Midazolam intravenous continusly infusion, Deep sedated (Ramsay 5)
  Other Names: Deep sedation
  Arms: Deep sedation
Drug: Light sedated — Midazolam intravenous continusly infusion, Light sedated (Ramsay 3)
  Other Names: Light sedation
  Arms: Light sedation

SUMMARY:
The acute respiratory distress syndrome (ARDS) is characterized by severe respiratory failure. Open Lung and Lung Protective Strategy have been proved to improve mortality of ARDS patients. Preserving spontaneous breathing (SB) is good for inflating the lung lobe near diaphram during mechanical ventilation, however, strong respiratory drive could generate more transpulmonary pressure in ARDS patients, which increase the stress and strain in injured lung. Nonetheless, it's not clear if sedative has any effects on transpulmonary pressure of ARDS patients.The purpose of this study is to investigate the effects of sedation on transpulmonary pressure of ARDS patients.

DETAILED DESCRIPTION:
Further study details as provided by Nanjing Zhong-da Hospital, School of Medicine, Southeast University

ELIGIBILITY:
Inclusion Criteria:

1. ARDS group patient (1) Acute onset of all of the following criteria within a 48-hour period:

   1. Requires positive pressure ventilation through an endotracheal tube
   2. Bilateral infiltrates consistent with edema on frontal chest radiograph, with a duration of no more than 7 days
   3. PaO2/FiO2 less than 300 while receiving positive end-expiratory pressure (PEEP) at more than 5 cm H2O for at least 4 hours, with a duration of no more than 7 days
   4. No clinical evidence of left atrial hypertension (2) Hemodynamics stable (dopamine <10ug/kg•min or norepinephrine <10ug/kg)
2. Surgical patient Surgical patient requires positive pressure ventilation through an endotracheal tube PaO2/FiO2 more than 300 Hemodynamics stable (dopamine <10ug/kg•min or norepinephrine <10ug/kg)

Exclusion Criteria:

* Age younger than 18 years or older than 85 years
* Cardiac failure
* Known pregnancy
* Increased intracranial pressure
* Severe neuromuscular disease
* Recent injury or other pathologic condition of the esophagus
* Pneumothorax
* Pleural effusion
* Diaphragmatic hernia
* Severe chronic respiratory disease
* End-stage chronic organ failure
* Expected survival of less than 24 hours
* Participation in another interventional study
* Attending physician declines to give consent for participant to enroll
* Patient or surrogate declines or is unable to give consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure generate by patient during deep or light sedation | 15 minutes during deep or light sedation
  Ispiratory transpulmonary pressure and expiratory transpulmonary pressure measured during sedation

SECONDARY OUTCOMES:
static compliance of respiratory system | 15min during deep or light sedation
  Crs measured during deep or light sedation
PaO2 | 15 minutes
  ABG after deep or light sedation

OTHER OUTCOMES:
MAP | 15 minutes
  MAP during deep or light sedation

CONTACTS AND LOCATIONS:
Overall Officials: Songqiao Liu, Doctor, Principal Investigator — Department of Critical Care Medicine, Nanjing Zhong-da Hospital, School of Medicine, Southeast University
Locations (1):
- Department of Critical Care Medicine, Nanjing Zhong-da Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No